CLINICAL TRIAL: NCT00049868
Title: Enhanced Linkage Maps From Family-Based Genetics Studies
Status: Completed | Type: Observational
Sponsor: Rutgers University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: Rutgers, The State University of New Jersey (Other)
Other Study IDs: 1203; R01HL071029 (NIH)
Record Dates: First submitted 2002-11-14; First posted 2002-11-15 (Estimated); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
To develop genetic maps for the genome-wide screening markers used by multiple investigators and to investigate map differences between sexes and different ethnic groups.

DETAILED DESCRIPTION:
BACKGROUND:

Meiotic linkage maps are the foundation of both linkage and linkage disequilibrium studies for mapping disease genes. Despite the importance of precise maps, existing genome-wide linkage maps were built using only a small collection of pedigrees, and so have wide confidence intervals surrounding estimates of map distance. Incorrect marker order and map distances can have a profound effect on linkage analyses. Using a sex-averaged map instead of a sex-specific map biases the lod scores upward, markedly increasing the false positive rate. Since it is very costly to follow-up many false-positive results, there is a clear need for more precise and accurate sex-specific genetic maps. Accurate estimates of meiotic map distance cannot be obtained by any means other than by linkage analysis using genotype data.

The study is in response to a Request for Applications entitled "NHLBI Innovative Research Grant Program" released in July, 2001. The purpose of the initiative is to support new approaches to heart, lung, and blood diseases and sleep disorders that use existing data sets or existing biological specimen collections whether obtained through National Heart, Lung, and Blood Institute support or not.

DESIGN NARRATIVE:

The genetic epidemiology study will build improved highly-precise sex-specific linkage maps utilizing thousands of individuals who have previously been genotyped. After filtering out obvious relationship and genotype errors, the study will incorporate methods that properly model for genotyping errors. In addition to creating precise maps for the scientific community, the study will also use these genotype data to study how recombination may vary between ethnic groups. The genotypes generated by the NHLBI Mammalian Genotyping Service are precisely the type of data required to produce more accurate maps. These data collections contain over 3,400 pedigrees with more than a 100-fold increase in information compared to that contained in the 8 CEPH families that have been used to construct current genome-wide linkage maps. The new maps will be made publicly available and the genotype data from the study will be accessible by the MAP-0-MAT linkage mapping server. In the future, the study will be broadened to incorporate genotype data from additional genotyping centers such as the Center for Inherited Disease Research (CIDR).

ELIGIBILITY:
No eligibility criteria

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2002-09; Study Completion 2005-08

CONTACTS AND LOCATIONS:
Overall Officials: Tara Matise — Rutgers, The State University of New Jersey